CLINICAL TRIAL: NCT06361277
Title: A Randomized, Open-label, Single Dose, Crossover Study to Compare the Pharmacokinetic Characteristics and Safety of JW0202 and C2202 or C2205 and JW0201 After Oral Administration in Healthy Volunteers
Brief Title: To Evaluate the Pharmacokinetic Characteristics and Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JW22104
Record Dates: First submitted 2024-03-27; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Treatment A: Co-administration of 2 tablets of C2205 and JW0201 Treatment B: Co-administration of 2 tablets of JW0202 and C2202
  Tablet, Oral, QD for 1 Day, Washout period is more than 21 days after administration
  Interventions: Drug: Reference Drug or Test Drug
- Group 2 (Other): Treatment A: Co-administration of 2 tablets of C2205 and JW0201 Treatment B: Co-administration of 2 tablets of JW0202 and C2202
  Tablet, Oral, QD for 1 Day, Washout period is more than 21 days after administration
  Interventions: Drug: Reference Drug or Test Drug

INTERVENTIONS:
Drug: Reference Drug or Test Drug — Tablet, Oral, QD for 1 Day, Washout period is more than 7 days after administration
  Other Names: Reference Drug(C2205 and JW0201) or Test Drug(JW0202 and C2202)

SUMMARY:
The objective is to evaluate the safety and pharmacokinetic characteristics after co-administration of JW0202 and C2202 and co-administration of C2205 and JW0201 in healthy volunteers under fasting conditions

DETAILED DESCRIPTION:
Pharmacokinetic characteristics: Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

Safety: All adverse events are summarized in terms of the number of subjects, expression rate, and number of expressions of adverse reactions by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the Inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
AUCt | Day1 0h ~ Day3 48h
  Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.
Cmax | Day1 0h ~ Day3 48h
  Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: MinGul Kim, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Clinical Trial Center, Jeonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No